CLINICAL TRIAL: NCT06302270
Title: Monitoring of Women and Children Exposed to the Combination of Elexacaftor-tezacaftor-ivacaftor During Bregnancy and Through Mother's Own Milk.
Brief Title: CFTR Modulators in Pregnancy and Postpartum
Status: Recruiting | Type: Observational
Sponsor: Region Stockholm (Other Government)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Other Study IDs: K2024-0507
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma and breastmilk
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- mother-infant dyads

SUMMARY:
Observational study on women with Cystic Fibrosis treated with CFTR modulators during pregnancy and postpartum and their children. Registration on maternal health parameters and effects of CFTR-modulators in the newborn infant as well as effects of exposure through mother's own milk.

ELIGIBILITY:
Inclusion Criteria:

Woman with cystic fibrosis who is pregnant and treated with Kaftrio. Newborn infant to the above mentioned woman

Exclusion Criteria:

none

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Woman with cystic fibrosis who is pregnant and treated with Kaftrio and her newborn infant
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2034-01-31 (Estimated); Study Completion 2039-01-31 (Estimated)

PRIMARY OUTCOMES:
Health effects in the newborn infant | 6 years

CONTACTS AND LOCATIONS:
Locations (1):
- Stockholm CF center, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
NO plan to share individual data. Not allowed.